CLINICAL TRIAL: NCT04450173
Title: A Phase II Trial of the Combination of Obinutuzumab, Ibrutinib, and Venetoclax in Patients With Previously Untreated Follicular Lymphoma
Brief Title: Obinutuzumab, Ibrutinib, and Venetoclax for the Treatment of Previously Untreated Stage II-IV Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pharmacyclics LLC. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#275; NCI-2020-01372 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#275 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2020-06-12; First posted 2020-06-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Ann Arbor Stage II Follicular Lymphoma; Ann Arbor Stage III Follicular Lymphoma; Ann Arbor Stage IV Follicular Lymphoma; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibrutinib; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (obinutuzumab, venetoclax, ibrutinib) (Experimental): Patients receive obinutuzumab IV over 60 minutes on days 1, 8, and 15 of cycle 1, day 1 of cycles 2-6, 8, 10, 12, 14, 16, 18, 20, 22, and 24. Patients also receive venetoclax PO QD on days 1-28 (days 4-28 of cycle 1) and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Biological: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well obinutuzumab, ibrutinib, and venetoclax work in treating patients with previously untreated stage II-IV follicular lymphoma. Immunotherapy with obinutuzumab may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Ibrutinib and venetoclax may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving obinutuzumab, ibrutinib, and venetoclax together may work better in treating follicular lymphoma compared to each drug alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of obinutuzumab combined with venetoclax and ibrutinib in patients with previously untreated follicular lymphoma (FL) (determined by a positron emission tomography [PET]/computed tomography [CT] complete response [CR] rate at 12 months as per International Workshop Lymphoma Response Criteria, Cheson 2014).

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of obinutuzumab in combination with venetoclax and ibrutinib in patients with untreated FL as assessed by frequency, severity, and relatedness of treatment-emergent adverse events (AEs) as well as frequency of treatment-emergent AEs requiring discontinuation or dose reduction of study drug.

II. To evaluate the efficacy of obinutuzumab in combination with venetoclax and ibrutinib in subjects with untreated FL as assessed by CR at 30 months, overall response rate (ORR) (CR + partial response [PR]), duration of response (DOR), time to next anti-lymphoma treatment (TTNT), progression-free survival (PFS), and OS.

OUTLINE:

Patients receive obinutuzumab intravenously (IV) over 60 minutes on days 1, 8, and 15 of cycle 1, day 1 of cycles 2-6, 8, 10, 12, 14, 16, 18, 20, 22, and 24. Patients also receive venetoclax orally (PO) once daily (QD) on days 1-28 (days 4-28 of cycle 1) and ibrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of follicular lymphoma (grades 1, 2, or 3a), untreated
* Able and willing to provide written informed consent and to comply with the study protocol
* Bi-dimensionally measurable disease, with at least one mass lesion >= 2 cm in longest diameter by CT, PET/CT, and/or magnetic resonance imaging (MRI)
* Must be in need of therapy as evidenced by at least one of the following criteria:

  * Bulky disease defined as:

    * A nodal or extranodal (except spleen) mass > 7 cm in its greater diameter or,
    * At least 3 nodal or extranodal sites >= 3 cm in diameter
  * Presence of at least one B symptom:

    * Fever (> 38 Celsius [C]) not due to infectious etiology
    * Night sweats
    * Weight loss > 10% in the past 6 months
  * Fatigue due to lymphoma
  * Splenomegaly (> 13 cm)
  * Compression syndrome (ureteral, orbital, gastrointestinal)
  * Any of the following cytopenias, due to lymphoma:

    * Hemoglobin =< 10 g/dL
    * Platelets =< 100 x 10^9/L
    * Absolute neutrophil count (ANC) < 1.5 x 10^9/L
  * Pleural or peritoneal effusion
  * Lactate dehydrogenase (LDH) > upper limit of normal (ULN) or beta (B)2 microglobulin > ULN
  * Other lymphoma-mediated symptoms as determined by the treating physician
* Stage II, III, or IV disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) > 1.0 x 10^9/L
* Platelet count > 50 x 10^9/L
* Prothrombin time (PT)/international normal ratio (INR) < 1.5 x (upper limit of normal) ULN and partial thromboplastin time (PTT) (activated partial thromboplastin time [aPTT]) < 1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder). When treated with warfarin or other vitamin K antagonists, then INR =< 3.0)
* Serum aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
* Creatinine clearance > 30 ml/min calculated by modified Cockcroft-Gault formula
* Bilirubin < 1.5 x ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin, in which case bilirubin should not exceed 3 g/dL
* Women of childbearing potential and men who are sexually active must practice reliable contraceptive measures started at least 4 weeks before study therapy and continued for 18 months following discontinuation of therapy. Females of childbearing potential must either completely abstain from heterosexual sexual contact or must use 2 methods of reliable contraception. Reliable contraceptive methods include 1 highly effective method (intrauterine device, birth control pills, hormonal patches, injections, vaginal rings, or implants) and at least 1 additional method (condom, diaphragm, or cervical cap) every time they have sex with a male. Males who are sexually active must be practicing complete abstinence or agree to a condom during sexual contact with a pregnant female or female of child bearing potential. Men must agree to not donate sperm during and for 90 days after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [B-hCG]) pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Known active central nervous system lymphoma or leptomeningeal disease
* Follicular lymphoma with evidence of diffuse large B-cell transformation
* Grade 3b follicular lymphoma
* Any prior history of other malignancy besides follicular lymphoma, unless the patient has been free of disease for >= 5 years and felt to be at low risk for recurrence by the treating physician, except:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (e.g., patients in whom dosing with obinutuzumab would be contraindicated for safety reasons)
* Known history of human immunodeficiency virus (HIV), active hepatitis C virus, active hepatitis B virus infection, or known bacterial, viral, fungal, mycobacterial, parasitic active systemic infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to the start of cycle 1

  * Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated
* Patients with a history of confirmed progressive multifocal leukoencephalopathy (PML), positive test results for human T-lymphotropic 1 virus, or suspected active or latent tuberculosis
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block. QT prolongation is not a significant ECG abnormality that would warrant exclusion
* Female subjects who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this study or within 90 days of last dose of study drug. Male subjects who plan to father a child while enrolled in this study or within 90 days after the last dose of study drug
* Administration of any investigational agent within 28 days of first dose of study drug
* Patients who have undergone major surgery within 14 days
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia)
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Subjects with chronic liver disease and hepatic impairment meeting Child-Pugh class C
* Subjects who received a strong cytochrome P450 (CYP) 3A4 inhibitor within 7 days prior to the first dose of ibrutinib or subjects who require continuous treatment with a strong CYP3A inhibitor or inducer
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | At 12 months
  Determined by positron emission tomography (PET)/computed tomography (CT) based on Cheson, Lugano classification 2014 as assessed by the investigator. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate.

SECONDARY OUTCOMES:
Frequency, severity, and relatedness of treatment-emergent adverse events (AEs) | Up to 30 days after completion of study treatment
  Adverse events will be graded and recorded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicity data by type and severity will be summarized by frequency tables.
Frequency of treatment-emergent AEs requiring discontinuation of study drug or dose reductions | Up to 30 days after completion of study treatment
  Adverse events will be graded and recorded according to NCI CTCAE version 5.0. Toxicity data by type and severity will be summarized by frequency tables.
CR rate | At 30 months (120 weeks)
  Determined by PET/CT based on Cheson, Lugano classification 2014 as assessed by the investigator. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate. The number and percentage of subjects with a CR will be tabulated.
Overall response rate (ORR) | Up to 2 years after completion of study treatment
  CR + partial response (PR), determined by PET/CT based on Cheson, Lugano classification 2014 as assessed by the investigator. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate. The number and percentage of subjects with an ORR will be tabulated. The best ORR will be recorded.
Duration of response | From the time by which measurement criteria for CR or PR, whichever is recorded first, is met until death or the first date by which progressive disease is documented, assessed up to 2 years after completion of study treatment
  CR + PR, determined by PET/CT based on Cheson, Lugano classification 2014 as assessed by the investigator. Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval (CI).
Time to next anti-lymphoma treatment | From the date of cycle 1/day 1 (each cycle is 28 days) to the date of first documented new anti-lymphoma treatment or death from any cause, assessed up to 2 years after completion of study treatment
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI. Comparison by important subgroups will be made using the log-rank test.
Progression-free survival | From the date of cycle 1/day 1 (each cycle is 28 days) to the date of first documented progression or death, assessed up to 2 years after completion of study treatment
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI. Comparison by important subgroups will be made using the log-rank test.
Overall survival | From the date of cycle 1/day 1 (each cycle is 28 days) to the date of death regardless of cause, assessed up to 2 years after completion of study treatment
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI. Comparison by important subgroups will be made using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — University of California, Davis
Locations (4):
- United States (4):
  - University of California, San Francisco (UCSF) Fresno, Fresno, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Diego, San Diego, California